CLINICAL TRIAL: NCT00558064
Title: Filtered Trial for Amlodipine Non-responder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Model: Parallel | Purpose: Treatment
Other Study IDs: 1235.13
Record Dates: First submitted 2007-10-29; First posted 2007-11-14 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan amlodipine combination; Amlodipine

INTERVENTIONS:
Drug: telmisartan+amlodipine
Drug: amlodipine

SUMMARY:
To demonstrate that a fixed-dose combination of telmisartan 40 mg plus amlodipine 5 mg is superior to amlodipine 5 mg alone in patients with essential hypertension and inadequately controlled with amlodipine 5 mg monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Essential hypertensive patients satisfying all of the following criteria;
2. Male or Female
3. Age > 20 years
4. Outpatient
5. Patients who are able to stop current anti-hypertensive therapy at Visit 1 if taking any anti-hypertensive medications
6. Patients with an ability to provide written informed consent in accordance with the related laws and guidelines such as Good Clinical Practice (GCP) and the Pharmaceutical Affairs Law.

Exclusion Criteria:

1. Taking four or more anti-hypertensive medications
2. Secondary hypertension
3. Mean seated diastolic blood pressure (DBP) > 114 mmHg and/or mean seated systolic blood pressure (SBP) > 200 mmHg at Visit 1, 2, 3, or 4, or mean seated DBP < 90 mmHg at Visit 3.
4. Sustained ventricular tachycardia or other clinically relevant cardiac arrhythmias
5. Congestive heart failure patients with the New York Heart Association (NYHA) functional class III-IV
6. History of myocardial infarction or cardiac surgery within last 6 months
7. History of coronary artery bypass graft or percutaneous coronary intervention (PCI) within last 3 months
8. History of unstable angina within last 3 months
9. Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of aortic or mitral valve
10. History of stroke or transient ischemic attack within last 6 months
11. History of sudden exacerbation of renal function with angiotensin II receptor blockers (ARBs) or angiotensin converting enzyme (ACE) inhibitors, or patients with post-renal transplant or post-nephrectomy
12. Experienced characteristic symptoms of angioedema during treatment with ARBs or ACE inhibitors
13. Known hypersensitivity to any component of the investigational drug , or a known hypersensitivity to dihydropyridine -derived drugs
14. Hepatic and/or renal dysfunction
15. Diagnosed biliary atresia or cholestasis
16. Hyperkalemia
17. Dehydration
18. Sodium deficiency
19. Chronic administration of high doses of acidic nonsteroidal anti-inflammatory drugs (NSAIDs)
20. Patients who cannot change to the restricted administration and dosage during study period
21. Pre-menopausal women who meet any one of the following 1 - 3:

    * Pregnant or possibly pregnant (1)
    * Nursing (2)
    * Desire to become pregnant during study period (3)
22. Drug or alcohol dependency
23. Complication of malignant tumour or a disease requiring immunosuppressants
24. Compliance of < 80% or > 120% during the run-in period
25. Receiving any investigational therapy within 3 months
26. Judged to be inappropriate by the investigator or the sub-investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2007-10; Primary Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (41):
- Japan (41):
  - 1235.13.037 Boehringer Ingelheim Investigational Site, Azumino, Nagano
  - 1235.13.023 Boehringer Ingelheim Investigational Site, Higashiosaka, Osaka
  - 1235.13.021 Boehringer Ingelheim Investigational Site, Itabashi-ku, Tokyo
  - 1235.13.014 Boehringer Ingelheim Investigational Site, Kashihara, Osaka
  - 1235.13.038 Boehringer Ingelheim Investigational Site, Kitaazumi-gun, Nagano
  - 1235.13.009 Boehringer Ingelheim Investigational Site, Kiyose, Tokyo
  - 1235.13.041 Boehringer Ingelheim Investigational Site, Kobe, Hyogo
  - 1235.13.035 Boehringer Ingelheim Investigational Site, Komoro, Nagano
  - 1235.13.003 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 1235.13.004 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 1235.13.027 Boehringer Ingelheim Investigational Site, Koriyama, Fukushima
  - 1235.13.007 Boehringer Ingelheim Investigational Site, Koshigaya, Saitama,
  - 1235.13.008 Boehringer Ingelheim Investigational Site, Koto-ku, Tokyo
  - 1235.13.005 Boehringer Ingelheim Investigational Site, Matsudo, Chiba
  - 1235.13.026 Boehringer Ingelheim Investigational Site, Mito, Ibaraki
  - 1235.13.013 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1235.13.016 Boehringer Ingelheim Investigational Site, Okayama, Okayama,
  - 1235.13.040 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1235.13.025 Boehringer Ingelheim Investigational Site, Saitama, Saitama
  - 1235.13.001 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1235.13.024 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1235.13.028 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1235.13.030 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1235.13.031 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1235.13.033 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1235.13.034 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1235.13.002 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1235.13.018 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1235.13.019 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1235.13.036 Boehringer Ingelheim Investigational Site, Shimoina-gun, Nagano
  - 1235.13.042 Boehringer Ingelheim Investigational Site, Shinjuku-ku, Tokyo
  - 1235.13.010 Boehringer Ingelheim Investigational Site, Shinjyuku-ku, Tokyo
  - 1235.13.011 Boehringer Ingelheim Investigational Site, Shinjyuku-ku,Tokyo
  - 1235.13.022 Boehringer Ingelheim Investigational Site, Shizuoka, Shizuoka
  - 1235.13.015 Boehringer Ingelheim Investigational Site, Suita, Osaka,
  - 1235.13.017 Boehringer Ingelheim Investigational Site, Takamatsu, Kagawa
  - 1235.13.029 Boehringer Ingelheim Investigational Site, Takamatsu, Kagawa
  - 1235.13.032 Boehringer Ingelheim Investigational Site, Takamatsu, Kagawa
  - 1235.13.012 Boehringer Ingelheim Investigational Site, Takaoka, Toyama
  - 1235.13.039 Boehringer Ingelheim Investigational Site, Takaoka,Toyama
  - 1235.13.020 Boehringer Ingelheim Investigational Site, Tsuchiura, Ibaraki

RESULTS

PARTICIPANT FLOW:
Groups:
- Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination: T40/A5 tablet, oral, once daily in the morning
- Amlodipine 5 mg Monotherapy: A5 capsule, oral, once daily in the morning
Period: Overall Study
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy
Started | 269 | 262
Completed | 264 | 257
Not Completed | 5 | 5
Not completed — Adverse Event | 3 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — No visit within allowance period | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy | Total
Number analyzed (Participants) | 269 | 262 | 531
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (9.6) | 56 (9.9) | 56.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 76 | 148
  Male | 197 | 186 | 383

OUTCOME MEASURES:

1. Primary Outcome: Reduction From Reference Baseline in Mean Seated Diastolic Blood Pressure at Trough (24-hour Post-dosing)
Description: The mean of the change value was least square mean which was calculated by analysis of covariance with factor treatment and center, and covariate baseline.
Time Frame: Baseline and 8 Weeks
Population: Full analysis set for blood pressure measurements, which was the analysis set including all the patients who had valid measurements at the reference baseline and at one or more time-points after the start of the double-blind maintenance period on final dose.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy
Number analyzed (Participants) | 263 | 257
mmHg | 9.56 (0.61) | 4.45 (0.61)
Statistical Analysis 1: Comparison: Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination vs Amlodipine 5 mg Monotherapy; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 5.11, 95% CI 2-sided [3.98 to 6.23], Standard Error of Mean 0.57 — Difference calculated as telmisartan 40 mg plus amlodipine 5 mg fixed-dose combination minus amlodipine 5 mg monotherapy

2. Secondary Outcome: Reduction From Reference Baseline in Mean Seated Systolic Blood Pressure at Trough (24-hour Post-dosing)
Description: as for outcome 1
Time Frame: Baseline and 8 Weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy
Number analyzed (Participants) | 263 | 257
mmHg | 13.04 (0.88) | 5.77 (0.88)

3. Secondary Outcome: Percentage of Patients With Seated Trough Diastolic Blood Pressure Less Than 90 mmHg at 8 Weeks (0 Percent at Baseline)
Description: Seated trough diastolic blood pressure defined as blood pressure in a sitting position no later than 24 hours after the last intake
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy
Number analyzed (Participants) | 263 | 257
percentage of patients | 68.1 | 47.1

4. Secondary Outcome: Percentage of Patients With Seated Trough Systolic Blood Pressure Less Than 140 mmHg at 8 Weeks (0 Percent at Baseline)
Description: Seated trough systolic blood pressure defined as blood pressure in a sitting position no later than 24 hours after the last intake
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy
Number analyzed (Participants) | 164 | 179
percentage of patients | 67.1 | 45.8

5. Secondary Outcome: Percentage of Patients Who Achieved an Adequate Response in Seated Trough Diastolic Blood Pressure at 8 Weeks (0 Percent at Baseline)
Description: Adequate response defined that seated trough diastolic blood pressure was <90 mmHg or decreased from reference baseline by >=10 mmHg at 8 weeks
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy
Number analyzed (Participants) | 263 | 257
percentage of patients | 74.5 | 50.2

6. Secondary Outcome: Percentage of Patients Who Achieved an Adequate Response in Seated Trough Systolic Blood Pressure at 8 Weeks
Description: Adequate response defined that seated trough systolic blood pressure was <140 mmHg or decreased from reference baseline by >=20 mmHg at 8 weeks (0 percent at baseline)
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy
Number analyzed (Participants) | 263 | 257
percentage of patients | 79.5 | 58.4

7. Secondary Outcome: Percentage of Patients With Optimal, Normal or High Normal Blood Pressure at 8 Weeks (0 Percent at Baseline)
Description: Optimal, normal, high normal blood pressure were defined as follows:
  * Optimal: Systolic blood pressure (SBP) < 120 mmHg and diastolic blood pressure (DBP) < 80 mmHg
  * Normal: SBP >= 120 mmHg or DBP >= 80 mmHg and SBP < 130 mmHg and DBP < 85 mmHg
  * High normal: SBP >= 130 mmHg or DBP >= 85 mmHg and SBP < 140 mmHg and DBP < 90 mmHg
  * No: SBP >= 140 mmHg and DPB >= 90 mmHg
Time Frame: 8 weeks
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy
Number analyzed (Participants) | 263 | 257
percentage of patients
  Optimal | 11.0 | 1.6
  Normal | 24.3 | 9.7
  High Normal | 26.6 | 23.0

8. Secondary Outcome: Clinically Relevant Abnormalities for Blood Chemistry, Pulse Rate, Laboratory Parameters and ECG
Description: Clinical relevant abnormalities for blood chemistry, pulse rate, laboratory parameters and ECG. New abnormal findings or worsening of baseline conditions were reported as Adverse Events.
Time Frame: First administration of randomised treatment to 24 hours post last dose of randomised treatment
Population: Treated set: Patients randomised to the double-blind treatment period who took at least one dose either of T40+A5 or A5 during the double-blind treatment period.
Measure: Number; unit: participants
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy
Number analyzed (Participants) | 269 | 262
participants
  Alanine aminotransferase increased | 1 | 0
  Aspartate aminotransferase increased | 1 | 0
  Blood creatine phosphokinase increased | 2 | 0
  Blood potassium increased | 0 | 1
  Blood urine present | 1 | 0
  Liver function test abnormal | 1 | 0
  Bradycardia | 1 | 0

ADVERSE EVENTS:
Time Frame: First administration of randomised treatment to 24 hours post last dose of randomised treatment
Arm/Group | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination | Amlodipine 5 mg Monotherapy
Serious Adverse Events (participants affected / at risk) | 1/269 | 2/262
Other Adverse Events (participants affected / at risk) | 25/269 | 34/262
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination (N=269) | Amlodipine 5 mg Monotherapy (N=262)
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Telmisartan 40 mg Plus Amlodipine 5 mg Fixed-dose Combination (N=269) | Amlodipine 5 mg Monotherapy (N=262)
Nasopharyngitis (Infections and infestations) | 25 | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract